CLINICAL TRIAL: NCT04775784
Title: Determination of SARS-Cov-2 Virus in Central Nervous System
Brief Title: Determination of COVID-19 Related Virus in Central Nervous System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Pietro Mortini, MD, Prof., Professor, IRCCS San Raffaele
Other Study IDs: NCH08-2020
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Testing; CNS Disease; CNS Infection
Keywords: SARS-Cov-2; CNS infection; Coronavirus; Brain
MeSH Terms: conditions — Central Nervous System Diseases; Central Nervous System Infections; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Brain tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult neurosurgical patients: Adult, both sex, neurosurgical patients candidate for intracranial surgery, able to sign informed consent.
  Interventions: Diagnostic Test: Determination of SARS-CoV2 presence in CNS

INTERVENTIONS:
Diagnostic Test: Determination of SARS-CoV2 presence in CNS — Brain tissue sampling

SUMMARY:
Coronavirus disease 2019 (COVID-19) is a highly infectious pandemic disease caused by SARS-CoV-2 virus. Central Nervous System (CNS) complications associated with COVID-19 might be secondary sequelae due to exuberant systemic innate-mediated hyper-inflammation, which may impair neurovascular endothelial function, disrupt blood brain barrier (BBB), activates CNS innate immune signaling pathways, and induces parainfectious autoimmunity, potentially contributing to the CNS manifestations. Although the predominant clinical manifestation of SARS-CoV-2 is characterized by dyspnea, unremitting fever and hypoxemic respiratory failure, neurologic manifestations do occur in most hospitalized SARS-CoV-2 patients and include non-specific encephalopathy, psychosis, meningitis/encephalitis, myelitis, cerebrovascular events, Guillain-Barre' syndrome, and cranial or peripheral neuropathies, such as anosmia and ageusia. To date, data about primary CNS involvement due to neurotropism and direct neuroinvasion are still lacking.

DETAILED DESCRIPTION:
Determination of SARS-CoV-2 presence in central nervous system

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patients candidate for CNS surgery
* Patients who have been tested for nasopharyngeal swab for SARS-CoV-2
* Patients who have been tested for serology test for anti SARS-CoV-2 immunoglobulinG (IgG) and immunoglobulinM (IgM) antibodies
* Patients able to sign informed consent

Exclusion Criteria:

* Patients not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients eligible to CNS surgery
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Determination of SARS-CoV-2 presence in the CNS | Surgery
  Brain tissue sampling analysis

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Mortini, MD, Prof., Principal Investigator — IRCCS San Raffaele Scientific Institute
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy

REFERENCES:
- [Background] Noorwali AA, Turkistani AM, Asiri SI, Trabulsi FA, Alwafi OM, Alzahrani SH, Rashid MM, Hegazy SA, Alzaydi MD, Bawakid KO. Descriptive epidemiology and characteristics of confirmed cases of Middle East respiratory syndrome coronavirus infection in the Makkah Region of Saudi Arabia, March to June 2014. Ann Saudi Med. 2015 May-Jun;35(3):203-9. doi: 10.5144/0256-4947.2015.203. PMID 26409794
- [Background] Montalvan V, Lee J, Bueso T, De Toledo J, Rivas K. Neurological manifestations of COVID-19 and other coronavirus infections: A systematic review. Clin Neurol Neurosurg. 2020 Jul;194:105921. doi: 10.1016/j.clineuro.2020.105921. Epub 2020 May 15. PMID 32422545
- [Background] Liotta EM, Batra A, Clark JR, Shlobin NA, Hoffman SC, Orban ZS, Koralnik IJ. Frequent neurologic manifestations and encephalopathy-associated morbidity in Covid-19 patients. Ann Clin Transl Neurol. 2020 Nov;7(11):2221-2230. doi: 10.1002/acn3.51210. Epub 2020 Oct 5. PMID 33016619
- [Background] Berger JR. COVID-19 and the nervous system. J Neurovirol. 2020 Apr;26(2):143-148. doi: 10.1007/s13365-020-00840-5. Epub 2020 May 23. PMID 32447630
- [Background] Najjar S, Najjar A, Chong DJ, Pramanik BK, Kirsch C, Kuzniecky RI, Pacia SV, Azhar S. Central nervous system complications associated with SARS-CoV-2 infection: integrative concepts of pathophysiology and case reports. J Neuroinflammation. 2020 Aug 6;17(1):231. doi: 10.1186/s12974-020-01896-0. PMID 32758257
- [Background] Liu J, Xie W, Wang Y, Xiong Y, Chen S, Han J, Wu Q. A comparative overview of COVID-19, MERS and SARS: Review article. Int J Surg. 2020 Sep;81:1-8. doi: 10.1016/j.ijsu.2020.07.032. Epub 2020 Jul 26. PMID 32730205
- [Background] Kumar A, Pareek V, Prasoon P, Faiq MA, Kumar P, Kumari C, Narayan RK. Possible routes of SARS-CoV-2 invasion in brain: In context of neurological symptoms in COVID-19 patients. J Neurosci Res. 2020 Dec;98(12):2376-2383. doi: 10.1002/jnr.24717. Epub 2020 Aug 31. PMID 32869376
- [Background] Song E, Zhang C, Israelow B, Lu-Culligan A, Prado AV, Skriabine S, Lu P, Weizman OE, Liu F, Dai Y, Szigeti-Buck K, Yasumoto Y, Wang G, Castaldi C, Heltke J, Ng E, Wheeler J, Alfajaro MM, Levavasseur E, Fontes B, Ravindra NG, Van Dijk D, Mane S, Gunel M, Ring A, Kazmi SAJ, Zhang K, Wilen CB, Horvath TL, Plu I, Haik S, Thomas JL, Louvi A, Farhadian SF, Huttner A, Seilhean D, Renier N, Bilguvar K, Iwasaki A. Neuroinvasion of SARS-CoV-2 in human and mouse brain. bioRxiv [Preprint]. 2020 Sep 8:2020.06.25.169946. doi: 10.1101/2020.06.25.169946. PMID 32935108
- [Background] Virhammar J, Kumlien E, Fallmar D, Frithiof R, Jackmann S, Skold MK, Kadir M, Frick J, Lindeberg J, Olivero-Reinius H, Ryttlefors M, Cunningham JL, Wikstrom J, Grabowska A, Bondeson K, Bergquist J, Zetterberg H, Rostami E. Acute necrotizing encephalopathy with SARS-CoV-2 RNA confirmed in cerebrospinal fluid. Neurology. 2020 Sep 8;95(10):445-449. doi: 10.1212/WNL.0000000000010250. Epub 2020 Jun 25. PMID 32586897
- [Background] Espindola OM, Brandao CO, Gomes YCP, Siqueira M, Soares CN, Lima MASD, Leite ACCB, Torezani G, Araujo AQC, Silva MTT. Cerebrospinal fluid findings in neurological diseases associated with COVID-19 and insights into mechanisms of disease development. Int J Infect Dis. 2021 Jan;102:155-162. doi: 10.1016/j.ijid.2020.10.044. Epub 2020 Oct 28. PMID 33127503
- [Background] Bernard-Valnet R, Pizzarotti B, Anichini A, Demars Y, Russo E, Schmidhauser M, Cerutti-Sola J, Rossetti AO, Du Pasquier R. Two patients with acute meningoencephalitis concomitant with SARS-CoV-2 infection. Eur J Neurol. 2020 Sep;27(9):e43-e44. doi: 10.1111/ene.14298. Epub 2020 May 30. No abstract available. PMID 32383343
- [Background] Paniz-Mondolfi A, Bryce C, Grimes Z, Gordon RE, Reidy J, Lednicky J, Sordillo EM, Fowkes M. Central nervous system involvement by severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2). J Med Virol. 2020 Jul;92(7):699-702. doi: 10.1002/jmv.25915. PMID 32314810
- [Background] Solomon IH, Normandin E, Bhattacharyya S, Mukerji SS, Keller K, Ali AS, Adams G, Hornick JL, Padera RF Jr, Sabeti P. Neuropathological Features of Covid-19. N Engl J Med. 2020 Sep 3;383(10):989-992. doi: 10.1056/NEJMc2019373. Epub 2020 Jun 12. No abstract available. PMID 32530583
- [Background] Pereira A. Long-Term Neurological Threats of COVID-19: A Call to Update the Thinking About the Outcomes of the Coronavirus Pandemic. Front Neurol. 2020 Apr 17;11:308. doi: 10.3389/fneur.2020.00308. eCollection 2020. No abstract available. PMID 32362868
- [Background] Yachou Y, El Idrissi A, Belapasov V, Ait Benali S. Neuroinvasion, neurotropic, and neuroinflammatory events of SARS-CoV-2: understanding the neurological manifestations in COVID-19 patients. Neurol Sci. 2020 Oct;41(10):2657-2669. doi: 10.1007/s10072-020-04575-3. Epub 2020 Jul 28. PMID 32725449